CLINICAL TRIAL: NCT06044610
Title: Utility of Transdermal Optical Imaging TOI) as a Non-invasive Measure of Hydration Status: Phase 3a for Model Development
Brief Title: Utility of Transdermal Optical Imaging (TOI) as a Non-invasive Measure of Hydration Status: Phase 3a for Model Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2306 3a
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Dehydration
Keywords: hydration; dehydration; euhydration; hypohydration; exercise; Transdermal Optical Imaging; TOI
MeSH Terms: conditions — Dehydration; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GENPOP passive dehydration (Experimental): 24-hour data collection using a parallel design comparison of TOI blood flow patterns vs. reference methods of hydration status in 10 PEP employees.
  Interventions: Other: GENPOP Passive dehydration (75% reduction in fluid intake
- EXERCISE without fluid replacement (Experimental): Randomized cross-over design in 15 moderately active non-employee participants. 90 minutes of standard cycling exercise trial in heat chamber. TOI signals will obtain blood flow patterns from the face to compare against reference methods of dehydration including body mass, urine specific gravity, urine color, and thirst.
  Interventions: Other: EXERCISE without fluid replacement
- GENPOP ad lib fluid intake (Other): 24-hour data collection using a parallel design comparison of TOI blood flow patterns vs. reference methods of hydration status in 10 PEP employees.
  Interventions: Other: GENPOP Ad lib fluid intake
- EXERCISE with fluid replacement (Other): Randomized cross-over design in 15 moderately active non-employee participants. 90 minutes of standard cycling exercise trial in heat chamber. TOI signals will obtain blood flow patterns from the face to compare against reference methods of dehydration including body mass, urine specific gravity, urine color, and thirst.
  Interventions: Other: EXERCISE with fluid replacement

INTERVENTIONS:
Other: GENPOP Passive dehydration (75% reduction in fluid intake — Over 24-hours
  Arms: GENPOP passive dehydration
Other: GENPOP Ad lib fluid intake — Over 24 hours
  Arms: GENPOP ad lib fluid intake
Other: EXERCISE without fluid replacement — 90-min standard cycling exercise trial in heat chamber
  Arms: EXERCISE without fluid replacement
Other: EXERCISE with fluid replacement — 90-min standard cycling exercise trial in heat chamber
  Arms: EXERCISE with fluid replacement

SUMMARY:
The primary objective of this study is to analyze smart phone-based Transdermal Optical Imaging (TOI) features to develop a model that can discern hypohydration from euhydration status including 1) a small feasibility study for 24-hour data collection in the general population using passive dehydration or ad libitum fluid intake (GENPOP), 2) an exercise study in moderately active participants in both dehydrated and euhydrated states (EXERCISE). TOI data will be collected alongside standard reference measures of hydration status.

This is an exploratory pilot proof of concept study with each subject serving as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* If female, subject is not pregnant
* For GENPOP study subject is 18-65 years of age, inclusive
* For EXERCISE study subject is 18-50 years of age, inclusive
* Subject is moderately-trained (engages in moderate-intensity, intermittent, or steady-state exercise at least 3 days per week for at least 1 hour at a time (EXERCISE session participants only)
* Subject does not smoke (or has quit for at least 6 months)
* Subject is not taking medication that may interfere with the study
* Subject has no health conditions that would prevent completion of the trial as indicated on the general health questionnaire (GHQ)
* Subject is willing to avoid alcohol consumption 24 hours prior to visit(s)
* Subject is willing to fast overnight (~8-12 hours)
* For GENPOP, subject is willing to refrain from vigorous exercise for 48 hours
* For EXERCISE, subject is willing to refrain from vigorous exercise for 24 hours prior to study visits
* Subject is willing to eat the exact same food the day prior to each visit to the laboratory
* Subject is willing to avoid wearing makeup to the study session
* Subject is willing to shave facial hair if predetermined during the informed consent session it will interfere with TOI measurement
* Able to speak, write, and read English
* Provision of written consent to participate

Exclusion Criteria:

* Subject has participated in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is allergic to alcohol or facial cleansing wipes
* Subject has a history of anaphylaxis or severe allergic reactions
* Subjects has a health condition or is taking medication that can be worsened by fluid restriction
* Subject has asthma or other condition which breathing can become labored during exercise (EXERCISE session participants only)
* Male subjects with a VO2max < 42 ml/kg/min and females with a VO2max < 38 ml/kg/min (EXERCISE session participants only)
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Transdermal optical imaging (TOI) signals | GENPOP: Before breakfast (~ 8 a.m.), before lunch ~11:30 a.m.), ~3:30 p,m., ~8.a.m. the following day. For EXERCISE, pre and post exercise session allowing for 30 minute cool down period.
  Blood flow patterns of the face obtained from the video camera on a smart phone
Standard measurements of hydration status | GENPOP: Before breakfast (~ 8 a.m.), before lunch ~11:30 a.m.), ~3:30 p,m., ~8.a.m. the following day. For EXERCISE, pre and post exercise sessions allowing for 30 minute cool down period.
  Body mass change, urine specific gravity, urine color (1-8 scale), and visual analogue scale to indicate thirst (1=not thirsty at all to 7 very, very thirsty)

SECONDARY OUTCOMES:
Demographics | At screening
  Age, sex, ethnicity, race
Fitzpatrick scale | At screening
  Classification of skin type 1 through 6, 1=White skin. Always burns, never tans, to 6=Black skin. Heavily pigmented. Never burns, tans very easily.
Mood scale | GENPOP: Before breakfast (~ 8 a.m.), before lunch ~11:30 a.m.), ~3:30 p,m., ~8.a.m. the following day
  9-point categorical scale from 1 (calm) to 9 (irritated)
Dietary and fluid intake | 24 hours prior to each visit through end of each study period.
  Log entries of food and drink
EXERCISE only: Rate of perceived exertion (RPE) | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  Borg scale (6-20 scale) from no exertion at all to maximal exertion
EXERCISE only: Heart rate | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  (beats/min)
EXERCISE only: Work rate | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  (watts, rpm)
EXERCISE only: Fluid intake (euhydrated state) | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  (fluid volume in milliliters)
EXERCISE only: Sweating rate | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  Rate of sweat over the course of the testing session.
EXERCISE only: Biomechanical and physiological features associated with dehydration, fatigue, and energy | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  Measured on staff iPad or iPhone to extract facial movements & voice quality features
EXERCISE only: Physical and mental energy | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  Rated from 1=Energetic to 6= Worn out and from 1=Never to 5=Always.
EXERCISE only: Grittiness score | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  8 item grit scale (examples: ideas, setbacks, goals)
EXERCISE only: Visual analogue scale for mental energy and fatigue | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  Marked on a horizontal line anchored by 0-100 mm with 0 (no energy and fatigue) to 100 mm (strongest feeling of energy and strongest feeling of fatigue ever felt)
EXERCISE only: Sweat biomarkers | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  (electrolyte and metabolites)
EXERCISE only: Saliva biomarkers | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  (osmolality and metabolites)
EXERCISE only: Fingertip capillary blood biomarkers | Two 90 minute standard cycling exercise trials separated by approximately 3 to 7 days
  (electrolytes and osmolality)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, PhD, Study Director — PepsiCo, Inc. Sports Science
Locations (2):
- United States (2):
  - PepsiCo R&D, Gatorade Sports Science Institute, Valhalla, New York
  - PepsiCo R&D, Gatorade Sports Science Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No